CLINICAL TRIAL: NCT04489069
Title: Multimodal and Multi-source Study of Developmental Psychopathology in Twin and Youth Cohorts: Integration of Neuroimaging, Neuropsychology and Gene-environment Measures
Brief Title: Developmental Psychopathology and the Gene-environment Interaction
Acronym: TwinAger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 212/2019-VERSIONE2
Record Dates: First submitted 2020-03-30; First posted 2020-07-28 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Developmental Psychological Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical, neuropsychological and MRI evaluations (Other)
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Clinical and Neuropsychological evaluations; Diagnostic Test: Drawing DNA sample

INTERVENTIONS:
Diagnostic Test: MRI — Magnetic Resonance Imaging (sturctural MRI, fMRI resting state and task related, DTI)
Diagnostic Test: Clinical and Neuropsychological evaluations — Clinical interviews and neuropsychological tests (paper/pencil and computer based)
Diagnostic Test: Drawing DNA sample — Saliva sample

SUMMARY:
The present is a followup study that aims at investigating the effect of genetic and environmental factors on the possible development of psychopathological conditions in a longitudinal perspective.

The final goal is to understand those factors that causing vulnerability to mental illness, eventually allowing better prevention and early detections of those persons with mental illness.

DETAILED DESCRIPTION:
The developmental psychopathology aims at studying the possible paths that psychiatric conditions may take from childhood, through adolescence till early adulthood. This developmental perspective has the final goal of allowing prevention and early detection of mental illness, which in turn should translate into better prognosis and outcomes.

Longitudinal research allows a better grasp on the illness etiology as it gives the opportunity of directly investigate the possible causal mechanisms and of defining the origins of psychopathological condition in adults.

Many factors of risk interact, across neurodevelopment, in determining the person's vulnerability to mental illness. For instance, temperament and psychopathological factors were proved to have a role. However, the existing knowledge is still fragmented and should be integrated by new knowledge on genetic and environmental factors. Thus, combining observations of neurodevelopment, as measured with neuro-imaging techniques at subsequent timepoints, with psychopathological and neuropsychological evaluations, as well as with detailed information on genetic, environmental and temperamental indexes, is crucial, as no similar exhaustive investigations are still available.

Furthermore, it must be bared in mind that the gene by environment interaction generates complex epigenetic effects on neurodevelopment, which should be monitored through a longer time lapse.

This topic has been studying this topic for years, by research groups with sites in Friuli Venezia Giulia and Bosisio Parini (Lecco, Lombardia), by mean of cross-sectional and longitudinal studies, involving samples of children and adolescents at risk of psychopathology and referred because of behavioral and/or emotional difficulties, experienced in the past or still ongoing. Also, the research involved a cohort of Twins recruited from the normal population and whose data would allow more fine tuned analyses of the bene by environment interaction.

In those first phases of study, instruments assessing the psychopathological risk were adapted to the Italian population and the associated cognitive marker were identified.

Also, some analysis investigated the effect of the environment on the psychopathological risk. Moreover, the influence of genetic factors is under now study, mainly focussing on epigenetic factors.

The research that is presented here is the followup of the previous investigations. In the previous year (2019) 33 participants underwent the follow up from the sample of children at psychopathological risk and who were chidden/adolescents at the time of the baseline evaluation.

During the current year the Twins cohort will be followed up. Half or more of the participants tested ad the baseline are expected to participate, which correspond to about 30 couples (60 participants). The subjects will undergo i) a magnetic resonance, including structural MRI, DTI, resting state fMRI, fMRI (during the fMRI sequences a concurrent task, tapping attention and emotional processes, is presented); ii) a psychopathological evaluation; iii) a self-rating evaluation, filling questionnaires measuring temperaments and assessing the possible presence of behavioral problems; iv) a neurocognitive evaluation; v) a drawing of biological-genetic sample (saliva).

ELIGIBILITY:
Inclusion Criteria:

* participants who already took part to the previous baseline evaluations carried out in our centers and signed consent to be contacted for future follow up

Exclusion Criteria:

* Current or previous neurological illness or trauma that involved the brain.
* Sensory impairments that can hamper the correct execution of the neurocognitive tasks and interviews.
* Intellectual disability (i.e. IQ<70 as estimated with the Wechsler Adult Intelligence Scale or the Wechsler Intelligence Scale for Children)

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance (MRI) of the Brain - MRI signal allowing tridimensional multiplanar reconstruction of the brain's structures | 10 minutes
  anatomical images obtained with high definition T1 weighted sequences of radio frequencies - the measure is a "signal (in Hz) to noise ratio" which is obtained from each voxel (tiny 3D portions of the brain)
MRI signal measuring the diffusion of weather particles across brain connections - Diffusion Tensor Imagning (DTI) | 10 minutes
  measures of the brain microstructure and connectivity - as in all MRI techniques, the measure is a "signal (in Hz) to noise ratio" which is obtained from each voxel (tiny 3D portions of the brain)
Functional Magnetic Resonance (fMRI) - MRI signal allowing to measure local brain's activity | 20 minutes
  BOLD signal reflecting the brain activity that is concurrent to the execution of the Continuous Performance Test associated to emotional stimuli, as well as at rest - as in all MRI techniques, the measure is a "signal (in Hz) to noise ratio" which is obtained from each voxel (tiny 3D portions of the brain)
clinical evaluation by mean of structures interviews - different interviews have different scales. In most of the cases the presence/absence of a psychiatric symptom is evaluated | 2 hours
  diagnosis or scores reflecting the degree of the presence or absence of a psychopathological condition or reflecting the personal temperament - The measures may vary on scales, for the most part the presence/absence (0-1) is recorded
neurocognitive evaluation - tests assessing general IQ, ability to produce words, drawing skills, attention's ability, memory. | 2 hours
  the output vary according to the test - they are accuracy scores (number of correct answers) or reaction times (milliseconds)
sample of saliva | >10 minutes for drawing the sample
  DNA single-nucleotide polymorphism from

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Bonivento, PhD, Principal Investigator — IRCCS E.Medea
Locations (1):
- IRCCS E.Medea, San Vito al Tagliamento, Pordenone, Italy

IPD SHARING:
Plan to Share IPD: No